CLINICAL TRIAL: NCT02512822
Title: Usefulness of Non-invasive Radiofrequency Therapy for Facial Contouring
Acronym: UNIRFFC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kangbuk Samsung Hospital (Other)
Collaborators: Cutera Inc. (Industry)
Responsible Party: Principal Investigator, Won-Serk Kim, Associate professor, Kangbuk Samsung Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: KBC13251D
Record Dates: First submitted 2015-07-27; First posted 2015-07-31 (Estimated); Last update posted 2015-07-31 (Estimated); Status verified 2015-07

CONDITIONS: Subcutaneous Fat
Keywords: radiofrequency; submental fat; fat reduction; body contouring

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Participants (Experimental): Noninvasive Radiofrequency
  Interventions: Procedure: Noninvasive Radiofrequency TruSculpt

INTERVENTIONS:
Procedure: Noninvasive Radiofrequency TruSculpt — Heating subcutaneous fat up to 45℃ continuously at least 3 minutes without surface damage and induces adipocytes apoptosis.
  Other Names: TruSculpt

SUMMARY:
To evaluate the efficacy of novel noninvasive RF technology for reduction of submental fat.

DETAILED DESCRIPTION:
Recently, Novel radiofrequency (RF) technology was introduced as a promising tool for non-invasive body and face contouring, which can heats subcutaneous fat up to 45℃ continuously without surface damage and induces adipocytes apoptosis.

Subjects with an excessive subcutaneous fat on the submental area received twice treatments at 1-month intervals. Clinical outcomes including the thickness of the submental fat (measured by ultrasound) and the submental circumference (measured by a tape measure), and clinical photographs were obtained at baseline, and 1-month and 6-month after last treatment.

ELIGIBILITY:
Inclusion Criteria:

* clinically appreciable localized excess of subcutaneous fat on the submental area
* no history of systemic underlying disease

Exclusion Criteria:

* any infectious or inflammatory skin diseases
* keloids
* psychiatric patients
* systemic underlying disease
* who had taken aesthetic procedure on the face, before 6-month

  * more than 5% weight change were dropped out.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Change from Baseline in thickness of the submental fat at 6 months | 6 months
  thickness of the submental fat measured by ultrasound
Change from Baseline in submental circumference at 6 months | 6 months
  thickness of the submental fat measured by a tape measure

SECONDARY OUTCOMES:
participants' assessment for improvement at 6 months | 6 months
  assessment for improvement by participants
participants' assessment for satisfaction at 6 months | 6 months
  assessment for satisfaction by participants

CONTACTS AND LOCATIONS:
Overall Officials: Won-Serk Kim, M.D., Ph.D., Study Director — Kangbuk Samsung Hospital

REFERENCES:
- [Background] Franco W, Kothare A, Ronan SJ, Grekin RC, McCalmont TH. Hyperthermic injury to adipocyte cells by selective heating of subcutaneous fat with a novel radiofrequency device: feasibility studies. Lasers Surg Med. 2010 Jul;42(5):361-70. doi: 10.1002/lsm.20925. PMID 20583242
- [Background] Franco W, Kothare A, Goldberg DJ. Controlled volumetric heating of subcutaneous adipose tissue using a novel radiofrequency technology. Lasers Surg Med. 2009 Dec;41(10):745-50. doi: 10.1002/lsm.20876. PMID 20014265